CLINICAL TRIAL: NCT06758479
Title: Correlations Between Disc Position and the Key Clinical Outcomes in TMD Patients: Cross-sectional Study
Brief Title: Differential Impact of TMJ Disc Displacement and Muscle Disorders on Pain, Function, and Quality of Life in TMD Patients
Acronym: DPTMD
Status: Completed | Type: Observational
Sponsor: King Khalid University (Other)
Collaborators: Rajiv Gandhi University of Health Sciences (Other)
Responsible Party: Principal Investigator, Sunil Kumar Vaddamanu, Dr, King Khalid University
Other Study IDs: ECC#2024-14; ECC#2024-14 (Other: Sri Rajiv Gandhi College of Dental Sciences & Hospital)
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Disorders (TMD); Disc Displacement; Functional Impairment
Keywords: Temporomandibular Joint Disorders (TMD); TMJ Disc Displacement; Jaw Pain and Dysfunction; MRI in TMD Assessment; Quality of Life in TMD; Helkimo Index; Oral Health Impact Profile (OHIP-14)
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Disc Position: Participants with an anatomically correct TMJ disc position as observed on MRI.
- Disc Displacement with Reduction (DDwR): Participants whose TMJ disc is displaced anteriorly at rest but returns to its normal position during mouth opening.
- Disc Displacement without Reduction (DDwoR): Participants whose TMJ disc remains displaced and does not return to its normal position during mouth opening

SUMMARY:
This study aims to explore the relationship between the position of the temporomandibular joint (TMJ) disc and key clinical outcomes in patients with temporomandibular disorders (TMD). TMD is a condition that can cause pain, difficulty in jaw movement, and reduced quality of life. The research examines how disc displacement, as seen on MRI scans, correlates with pain levels, jaw function, and overall well-being. By better understanding these connections, the study seeks to provide insights that could improve the diagnosis and management of TMD, enhancing patient care and outcomes. This observational study involves non-invasive clinical and imaging assessments of TMD patients.

DETAILED DESCRIPTION:
This observational, cross-sectional study investigates the correlation between temporomandibular joint (TMJ) disc position and clinical outcomes in patients diagnosed with temporomandibular disorders (TMD). TMD encompasses conditions causing pain, jaw dysfunction, and diminished quality of life. The study evaluates disc displacement using magnetic resonance imaging (MRI) and measures clinical outcomes such as pain severity (Visual Analog Scale), functional limitations (Helkimo Index), and quality of life (Oral Health Impact Profile-14).

Participants include 100 individuals aged 18-65 with clinically confirmed TMD. Data collection involves clinical evaluations and MRI imaging to classify disc displacement into categories such as normal, with reduction, and without reduction. Statistical analyses, including correlation and regression, identify relationships between disc position and outcomes while accounting for confounding factors.

The findings aim to improve understanding of the pathophysiology of TMD and guide diagnostic and therapeutic strategies for better patient outcomes. The study adheres to ethical guidelines, ensuring informed consent and patient confidentiality.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18 and 65 years.
2. Diagnosed with temporomandibular disorders (TMD) based on clinical examination and imaging (MRI).
3. Presence of at least one of the following symptoms:

   * Jaw pain
   * Restricted jaw movement
   * Clicking sounds in the temporomandibular joint (TMJ)
4. No history of recent jaw or facial trauma.
5. No systemic diseases affecting the TMJ or musculoskeletal system (e.g., rheumatoid arthritis).
6. Able to provide informed consent.

Exclusion Criteria:

1. History of major jaw or facial trauma within the last six months.
2. Systemic conditions that might affect TMJ function, such as autoimmune diseases or bone disorders.
3. Previous TMJ surgery or other major interventions.
4. Pregnant or lactating women.
5. Inability to undergo MRI due to contraindications (e.g., metal implants, pacemakers).
6. Severe malocclusion or other dental/medical conditions interfering with TMD diagnosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 to 65 years diagnosed with temporomandibular disorders (TMD). Participants are recruited from a multidisciplinary clinic specializing in TMD diagnosis and management. Eligible individuals present with clinical symptoms such as jaw pain, restricted movement, or clicking sounds in the temporomandibular joint (TMJ) and have their diagnosis confirmed through physical examination and MRI imaging. The study excludes individuals with systemic diseases affecting the TMJ, recent jaw trauma, prior TMJ surgeries, and conditions that may interfere with TMD diagnosis or imaging. The population is representative of patients seeking care for TMD, allowing for analysis of clinical and imaging correlations.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-12-26 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Measured at the time of enrollment.
  Pain severity will be assessed using the Visual Analog Scale (VAS), with scores ranging from 0 (no pain) to 10 (worst possible pain)
Pain Severity | Measured at the time of enrollment.
  Pain severity will be assessed using the Visual Analog Scale (VAS), but focused on the patient's retrospective assessment of the worst pain experienced within the last week.
Pain Severity | Measured at the time of enrollment.
  Pain severity will be assessed using the Visual Analog Scale (VAS), considering the patient's average pain experienced over the past month.

SECONDARY OUTCOMES:
Functional Limitations | Measured at the time of enrollment
  Functional limitations will be evaluated using the Helkimo Index, assessing parameters such as jaw movement and mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K Vaddamanu, MDS, Principal Investigator — snu@kku.edu.sa
Locations (1):
- Sri Rajiv Gandhi College of Dental Sciences & Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared because the study involves sensitive patient information, including clinical and imaging data, which are subject to strict privacy and confidentiality regulations. Additionally, the scope of the study does not include provisions for external data sharing, as the data is intended solely for the purposes of this research and its analysis. Access to the data is restricted to the research team to ensure compliance with ethical standards and institutional review board (IRB) requirements.